CLINICAL TRIAL: NCT01827098
Title: A Randomized Controlled Clinical Trial of Regenerative Protocols to Treat Immature Necrotic Teeth
Brief Title: A Clinical Study to Compare Two Revascularization Protocols to Treat Non-vital Teeth With Incomplete Root Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Tatiana Botero, Clinical Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM-00066353
Record Dates: First submitted 2013-01-07; First posted 2013-04-09 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Dental Pulp Necrosis; Disorder of Tooth Development
Keywords: Immature teeth; Calcium Hydroxide; Blood clot; Revascularization; Revitalization
MeSH Terms: conditions — Dental Pulp Necrosis; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed induction (Experimental): The root canal is disinfected and calcium hydroxide is placed in the canal. Blood clot is induced in the canal 4 weeks later. Endodontic Regeneration is performed.
  Interventions: Procedure: Endodontic Regeneration
- Immediate Induction (Experimental): Blood clot is induced after disinfection of the canal during the same visit. Endodontic regeneration is performed.
  Interventions: Procedure: Endodontic Regeneration

INTERVENTIONS:
Procedure: Endodontic Regeneration — Blood clot formation is induced in the root canal after disinfection. Collagen material is placed over the clot. The canal access is sealed with white MTA and glass ionomer restoration. Permanent restoration is placed 3 months later on top of the MTA.

SUMMARY:
Both methods tested in this study disinfect the non-vital root canals and induce blood clot formation inside the root canal. One method places calcium hydroxide inside the root canal after disinfection and the blood clot is induced four weeks later.

The other method performs disinfection and induction of blood clot in one appointment. The investigators hypothesize that both methods will obtain the same success rate in eliminating infection, increase in root length and canal walls thickness.

DETAILED DESCRIPTION:
Collagen is placed on top of the blood clot, followed by white MTA. Glass ionomer is used to seal the access to the canal, which will be replaced by a permanent restoration 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or having a mild systemic disease (ASA Physical Status 1 or 2), with no contraindications to the treatment.
* Cooperative.
* Clinical diagnosis of pulp necrosis based on cold test, electric pulp test as well as an identified cause of pulp necrosis such as caries, deep restorations, dental anomalies, history of trauma, associated with radiographic and/or clinic signs of periapical lesion.
* Open apex with a diameter of at least 1mm. For teeth with more than one apical foramen, at least one foramen needs to be 1mm wide.
* Tooth is restorable and periodontally stable.

Exclusion Criteria:

* Pregnancy.
* Evidence of pathological external or internal root resorption, root fracture or ankylosis.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Absence of infection and inflammation. | 12 and 24 months after the induction of blood clot
  clinic evaluation to determine the status of periodontal tissues

SECONDARY OUTCOMES:
Changes in root length and canal wall width | Baseline and 12 months after the induction of blood clot
  Radiographic evaluation of these changes at 12 m as compared to the initial x-rays
Changes in root length and canal wall width | Baseline and 24 months after the induction of blood clot
  Radiographic evaluation of these changes at 24 m as compared to the initial x-rays

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana M Botero, DDS, MS, Principal Investigator — University of Michigan
Locations (1):
- Graduate Endodontic Clinic, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Banchs F, Trope M. Revascularization of immature permanent teeth with apical periodontitis: new treatment protocol? J Endod. 2004 Apr;30(4):196-200. doi: 10.1097/00004770-200404000-00003. PMID 15085044
- [Background] Thibodeau B, Trope M. Pulp revascularization of a necrotic infected immature permanent tooth: case report and review of the literature. Pediatr Dent. 2007 Jan-Feb;29(1):47-50. PMID 18041512
- [Background] Hargreaves KM, Geisler T, Henry M, Wang Y. Regeneration potential of the young permanent tooth: what does the future hold? Pediatr Dent. 2008 May-Jun;30(3):253-60. PMID 18615992
- [Background] Botero TM, Tang X, Gardner R, Hu JCC, Boynton JR, Holland GR. Clinical Evidence for Regenerative Endodontic Procedures: Immediate versus Delayed Induction? J Endod. 2017 Sep;43(9S):S75-S81. doi: 10.1016/j.joen.2017.07.009. PMID 28844307
- [Background] Rosa V, Botero TM, Nor JE. Regenerative endodontics in light of the stem cell paradigm. Int Dent J. 2011 Aug;61 Suppl 1(Suppl 1):23-8. doi: 10.1111/j.1875-595X.2011.00026.x. PMID 21726222
- [Background] Schneider R, Holland GR, Chiego D Jr, Hu JC, Nor JE, Botero TM. White mineral trioxide aggregate induces migration and proliferation of stem cells from the apical papilla. J Endod. 2014 Jul;40(7):931-6. doi: 10.1016/j.joen.2013.11.021. Epub 2014 Jan 16. PMID 24935538
- [Background] Botero TM, Son JS, Vodopyanov D, Hasegawa M, Shelburne CE, Nor JE. MAPK signaling is required for LPS-induced VEGF in pulp stem cells. J Dent Res. 2010 Mar;89(3):264-9. doi: 10.1177/0022034509357556. Epub 2010 Jan 28. PMID 20110511
- See also: American Association of Endodontics - Considerations for Regenerative Procedures — http://www.aae.org/regeneration/